CLINICAL TRIAL: NCT03756805
Title: Selective Upper Airway Stimulation Compared to Continuous Positive Airway Pressure Therapy in Patients With Obstructive Sleep Apnea: a Prospective Cohort Study
Brief Title: Upper Airway Stimulation Versus Continuous Positive Airway Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAS vs. CPAP
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; hypoglossal nerve stimulation; upper airway stimulation; surgical treatment sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Patients with moderate to severe sleep apnea (apnea-hypopnea index (AHI) between 15 / h and 65 / h) are included in the period 2014-2018. The patients are assigned to two groups: group 1, who are receiving PAP therapy and group 2, who are receiving upper airway stimulation. All patients receive polysomnography (PSG) in the sleep laboratory prior to therapy and are followed up on average 12 months after initiation of therapy by PSG or a home sleep test. This protocol is close to the daily clinical routine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (CPAP) (Active Comparator): Patient, who are receiving a CPAP
  Interventions: Device: continuous positive airway pressure
- Group 2 (UAS) (Experimental): Patient, who are receiving a device for upper airway stimulation
  Interventions: Device: upper airway stimulation

INTERVENTIONS:
Device: upper airway stimulation — One group of patients with UAS
  Other Names: Inspire
  Arms: Group 2 (UAS)
Device: continuous positive airway pressure — One group of patients with CPAP
  Arms: Group 1 (CPAP)

SUMMARY:
Standard therapy in patients with obstructive sleep apnea (OSA) is continuous positive airway pressure (CPAP). 30% to 50% are not adherent to this therapy and need an alternative treatment. Hypoglossal nerve stimulation or selective upper airway stimulation has been developed since several years. The aim of this clinical trial is to compare both treatments with each other.

DETAILED DESCRIPTION:
6% to 13% of the western industrialized population suffer from obstructive sleep apnea (OSA). During sleep in the pharyngeal airway a relaxation of the muscles occurs with increasing depth of sleep. Finally, this relaxation, due to the anatomical conditions, lead to obstructions of the respiratory tract, resulting in respiratory arrest (apnea) and minor respiratory changes such as hypopneas or flow limitations. The symptoms of this disease manifest themselves with varying degrees. Increased daytime sleepiness, snoring, and increased risk of cardiovascular disease can result. A significant reduction in overall quality of life can be associated with OSAS. The gold standard treatment for obstructive sleep apnea is CPAP (continuous positive airway pressure). But only about 50% to 70% of patients continue to use their device after 2 years of initial CPAP therapy. This means that 30% to 50% of patients are no longer cared for their obstructive sleep apnea. A certain proportion of younger patients, in particular, reject nocturnal ventilation therapy with CPAP from the beginning. For these patients selective upper airway stimulation (UAS) is a therapy option.

Therefore the patient receives surgically a subcutaneous stimulation device under the clavicle, which receives a signal from a respiratory sensor to selectively stimulate the hypoglossal nerve. The respiratory sensor is located in the 4th or 5th intercostal space between the patient's external and internal rib muscles. This can be used to record the patient's breathing, which allows a matched stimulation of the hypoglossal nerve. The actual stimulation lead is attached to the medial branches of the hypoglossal nerve, which are responsible for the protrusion of the tongue, in order to enable appropriate stimulation.

In this prospective cohort study, selective upper airway stimulation (UAS) will now be compared with CPAP therapy. Patients receiving CPAP therapy are compared to UAS patients who receive an upper airway stimulation. Both methods are procedures established in clinical routine, and during this investigation, the general clinical course is not deviated. Randomization does not occur because CPAP therapy is a conservative therapy and UAS therapy is a surgical therapy. Furthermore, for UAS therapy, there must be a CPAP incompliance, so that a surgical concept is justified. The CPAP group should comply with the body mass index and age of the UAS group.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who either received UAS implantation (Inspire therapy) in our Department of Otorhinolaryngology, Head and Neck Surgery at the Klinikum rechts der Isar and all patients who received a CPAP therapy since July 2013, are invited to participate in this clinical examination.

Exclusion Criteria:

* patients with the age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
AHI | reduction from baseline to 12 months
  Apnea Hypopnea Index measured in events per hour
ODI | reduction from baseline to 12 months
  Oxygen desaturation index measured in events per hour

SECONDARY OUTCOMES:
ESS | improvement from baseline to 12 months
  Epworth Sleepiness Scale
FOSQ | improvement from baseline to 12 months
  Functional Outcome of Sleep Questionnaire
Usage | usage hours per night at 12 months
  Usage Hour per Night

CONTACTS AND LOCATIONS:
Locations (1):
- Technical University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heiser C, Steffen A, Strollo PJ Jr, Giaie-Miniet C, Vanderveken OM, Hofauer B. Hypoglossal nerve stimulation versus positive airway pressure therapy for obstructive sleep apnea. Sleep Breath. 2023 May;27(2):693-701. doi: 10.1007/s11325-022-02663-6. Epub 2022 Jul 2. PMID 35779166
- See also: Official Website of the Department — http://www.schlaf-hno.de